CLINICAL TRIAL: NCT06159790
Title: A Randomized, Double-blind, Parallel-group Study to Compare Efficacy, Safety, and Immunogenicity of GME751 (Proposed Pembrolizumab Biosimilar) and EU-authorized Keytruda® in Adult Participants With Untreated Metastatic Non-squamous Non-small Cell Lung Cancer (NSCLC)
Brief Title: A Study to Compare Efficacy, Safety, and Immunogenicity of GME751 and EU-authorized Keytruda in Adult Participants With Untreated Metastatic Non-squamous Non-small Cell Lung Cancer (NSCLC)
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: In light of the evolving regulatory landscape and growing indications that major Health Authorities will move towards a streamlined clinical development, Sandoz took a strategic decision and is minimizing its CGME751A12301 clinical study.
Sponsor: Sandoz (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CGME751A12301
Record Dates: First submitted 2023-10-10; First posted 2023-12-07 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Metastatic NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GME751 + pemetrexed + carboplatin or cisplatin (Experimental): Participants will receive GME751 + pemetrexed + carboplatin or cisplatin via intravenous (IV) infusion.
  Interventions: Drug: GME751
- Keytruda-EU + pemetrexed + carboplatin or cisplatin (Active Comparator): Participants will receive Keytruda-EU + pemetrexed + carboplatin or cisplatin via intravenous (IV) infusion.
  Interventions: Drug: Keytruda-EU

INTERVENTIONS:
Drug: GME751 — Drug: GME751 Concentrate for solution for infusion, Biologic, Liquid in vial, 100 mg, 200 mg every 3 weeks, i.v. infusion Drug: Pemetrexed (i.v. infusion) Drug: Carboplatin or Cisplatin (i.v. infusion)
  Arms: GME751 + pemetrexed + carboplatin or cisplatin
Drug: Keytruda-EU — Drug: Keytruda-EU Concentrate for solution for infusion, biologic, liquid in vial, 100 mg, 200mg every 3 weeks, i.v. infusion Drug: Pemetrexed (i.v. infusion) Drug: Carboplatin or Cisplatin (i.v. infusion)
  Arms: Keytruda-EU + pemetrexed + carboplatin or cisplatin

SUMMARY:
The purpose of this study is to investigate the efficacy, safety, and immunogenicity of GME751 compared with Keytruda® (pembrolizumab) in participants with untreated metastatic non-squamous NSCLC (irrespective of PD-L1 status), without sensitizing EGFR or ALK mutations.

DETAILED DESCRIPTION:
Eligible participants will be randomized in a 1:1 ratio to receive either GME751, or European Union (EU)-authorized pembrolizumab (Keytruda-EU) in combination with chemotherapy. The maximum study duration for a participant will be approximately 56 weeks including screening.

Treatment duration is 52 weeks (17 treatment cycles of study treatment GME751 or Keytruda-EU in combination with chemotherapy, each cycle with a duration of 3 weeks).

Participants will discontinue study participation in case of disease progression, unacceptable toxicity or other reasons.

Participants who are benefiting from treatment with pembrolizumab without signs of progression or unacceptable toxicity will be eligible for continued pembrolizumab treatment via most suitable option based on the respective country regulations.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Untreated metastatic NSCLC
* Absence of tumor activating EGFR mutations and absence of ALK gene rearrangements
* Measurable disease according to RECIST 1.1
* Adequate organ function
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1

Exclusion Criteria:

* Squamous cell or mixed histology in NSCLC
* Known history of hypersensitivity (grade ≥3) to pembrolizumab, chemotherapy or their excipients
* Active autoimmune disease that has required chronic systemic treatment in the past 2 years.
* Received live vaccine ≤30 days before the first study treatment
* Prior treatment with pembrolizumab or any other anti-PD-1, or anti-PD-L1 or anti-PD-L2, or anti-CTLA-4 agent or any antibody targeting other immune-regulatory receptors or mechanisms for lung cancer.

Other protocol-defined inclusion/exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2024-04-29 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Best Overall Response (BOR) | up to 9 months from date of randomization
  Best Overall Response (BOR) of either Complete Response (CR) or Partial Response (PR) up to 9 months according to RECIST 1.1 as assessed by Blinded Central Imaging

CONTACTS AND LOCATIONS:
Locations (60):
- Sandoz Investigational Site, Fountain Valley, California, United States
- Bosnia and Herzegovina (3):
  - Sandoz Investigational Site, Banja Luka
  - Sandoz Investigational Site, Sarajevo
  - Sandoz Investigational Site, Zenica
- Brazil (5):
  - Sandoz Investigational Site, Belo Horizonte
  - Sandoz Investigational Site, Fortaleza
  - Sandoz Investigational Site, Ipatinga
  - Sandoz Investigational Site, Porto Alegre
  - Sandoz Investigational Site, São José do Rio Preto
- Georgia (2):
  - Sandoz Investigational Site, Batumi
  - Sandoz Investigational Site, Tbilisi
- Sandoz Investigational Site, Rosenheim, Germany
- India (8):
  - Sandoz Investigational Site, Ahmedabad
  - Sandoz Investigational Site, Bhubaneswar
  - Sandoz Investigational Site, Hyderabad
  - Sandoz Investigational Site, Mumbai
  - Sandoz Investigational Site, Nagpur
  - Sandoz Investigational Site, Nashik
  - Sandoz Investigational Site, New Delhi
  - Sandoz Investigational Site, Varanasi
- Japan (7):
  - Sandoz Investigational Site, Asahikawa
  - Sandoz Investigational Site, Funabashi
  - Sandoz Investigational Site, Hiroshima
  - Sandoz Investigational Site, Kanazawa
  - Sandoz Investigational Site, Niigata
  - Sandoz Investigational Site, Okayama
  - Sandoz Investigational Site, Sapporo
- Malaysia (7):
  - Sandoz Investigational Site, Johor Bahru
  - Sandoz Investigational Site, Kuala Lumpur
  - Sandoz Investigational Site, Kuantan
  - Sandoz Investigational Site, Kuching
  - Sandoz Investigational Site, Malacca
  - Sandoz Investigational Site, Petaling Jaya
  - Sandoz Investigational Site, Putrajaya
- Philippines (3):
  - Sandoz Investigational Site, Bacolod
  - Sandoz Investigational Site, Cebu City
  - Sandoz Investigational Site, Makati
- Romania (2):
  - Sandoz Investigational Site, Cluj-Napoca
  - Sandoz Investigational Site, Floreşti
- Sandoz Investigational Site, Kragujevac, Serbia
- Spain (4):
  - Sandoz Investigational Site, A Coruña
  - Sandoz Investigational Site, Córdoba
  - Sandoz Investigational Site, Madrid
  - Sandoz Investigational Site, Oviedo
- Taiwan (4):
  - Sandoz Investigational Site, Douliu
  - Sandoz Investigational Site, Kaohsiung City
  - Sandoz Investigational Site, Taichung
  - Sandoz Investigational Site, Taipei
- Thailand (2):
  - Sandoz Investigational Site, Bangkok
  - Sandoz Investigational Site, Khon Kaen
- Turkey (Türkiye) (7):
  - Sandoz Investigational Site, Adana
  - Sandoz Investigational Site, Bursa
  - Sandoz Investigational Site, Gaziantep
  - Sandoz Investigational Site, Istanbul
  - Sandoz Investigational Site, Malatya
  - Sandoz Investigational Site, Sakarya
  - Sandoz Investigational Site, Yüreğir
- Vietnam (3):
  - Sandoz Investigational Site, Hanoi
  - Sandoz Investigational Site, Hà Nội
  - Sandoz Investigational Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: No